CLINICAL TRIAL: NCT01754584
Title: The Effect and Mechanism of Hyaluronan on the Mucociliary Differentiation of Human Respiratory Epithelial Cells
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Far Eastern Memorial Hospital-IRB, Far Eastern Memorial Hospital-IRB
Other Study IDs: FEMH 97055
Record Dates: First submitted 2009-02-06; First posted 2012-12-21 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-11

CONDITIONS: Respiratory System Defect
Keywords: hyaluronan including concentrations; molecular weight; mucociliary differentiation; human respiratory epithelial cells

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The mucociliary system of nasal mucosa, which is composed of the ciliated respiratory epithelium, the mucous blanket, and the mucus-producing glands, is an important defense component of the respiratory system. Therefore, it is important to maintain intact inner respiratory mucociliary epithelium in reconstruction of large respiratory defect and in the development of tissue engineering trachea. Hyaluronan derivatives, which are biodegradable and non-immunogenic, have already proved to be effective as a scaffold for chondrocytes. However, the feasibility of use as a scaffold for respiratory epithelial cells remained unexplored. The aim of the study is to investigate the effect of hyaluronan including concentrations and molecular weight on the mucociliary differentiation of human respiratory epithelial cells (HREC). If hyaluronan is able to promote mucociliary differentiation of HREC, the investigators can synthesize hyaluronan derivatives serving as ideal biomaterials for respiratory tissue engineering and tissue-engineered trachea in the future.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS UNDERWENT SEPTOMEATOPLASTY

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: PATIENTS UNDERWENT SEPTOMEATOPLASTY
Sampling Method: Non-Probability Sample
Dates: Start 2009-01